CLINICAL TRIAL: NCT05022095
Title: "Validated Language Transfer of the Spinal Cord Injury-Spasticity Evaluation Tool to German Language"
Acronym: SCI-SETde
Status: Completed | Type: Observational
Sponsor: Swiss Paraplegic Research, Nottwil (Network)
Responsible Party: Principal Investigator, Tim Reck, Head of Interventional/Conservative pain medicine, Swiss Paraplegic Research, Nottwil
Other Study IDs: 2021-05
Record Dates: First submitted 2021-08-16; First posted 2021-08-26 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: SCI - Spinal Cord Injury; Spastic
Keywords: Spasticity; Spinal Cord Injury; Activities of daily living; Quality of Life
MeSH Terms: conditions — Spinal Cord Injuries; Muscle Spasticity | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SCI Patients with ongoing spasticity: SCI Patients that are either seen in clinical routine due to fillings or controls of their intrathecal injection pumps or stationary patients will be informed about the project, they are granted with enough time to decide whether they want participate or not. After giving Informed Consent they will be administered a set of questionnaires including SCI-SETde, PSFS (adapted to german), SCIM-SR in german as well as self-evaluation of spasticity severity and intensity. The SCI-SETde will be filled in again one week later to evaluate test-retest reliability. Overall, the burden for the patients is kept at minimum. There are no expected risks or harm to the patients.
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — Diverse questionnaires have to be filled in.

SUMMARY:
To better depict the full range of spasticity after Spinal Cord Injury (SCI) there is a need to take into account the patients perspective and their experiences during daily life. In 2007 the Spinal Cord Injury-Spasticity Evaluation Tool (SCI-SET) was created and validated. This specific questionnaire addresses the influence of spasticity on the daily life of SCI patients and takes into account negative as well as positive effects of spasticity to fulfill certain tasks. Until now this questionnaire is only available in english, turkish and persian language. Therefore, the investigators translated and culturally adapted this questionnaire and within this study this questionnaire shall be validated in a small cohort of SCI patients. The patients will fill in several different questionnaires at a first meeting and one week later the SCI-SETde questionnaire again to evaluate test-retest properties. Recruiting will happen completely at the Swiss Paraplegic Centre Nottwil, Switzerland.

DETAILED DESCRIPTION:
Life expectancy of persons in the acute phase after a spinal cord injury (SCI) dramatically increased in the second half of the last century. The long-term mortality (more than two years post-injury) is still an issue and a strong contributing risk factor are secondary health conditions also including spasticity. Spasticity has been reported to be present in 74% of people in a recent cross-sectional study investigating a cohort including Swiss residents. There are many different forms of spasticity seen in patients as well as varying definitions found in the literature. Furthermore it is recognized that spasticity may have both negative as well as positive impacts on daily life.

Spasticity should not solely be assessed with objective measures and the inclusion of the patient's perspective and personal perception is crucial to completely address and trace out spasticity in each individual. The patient reported impact of spasticity measure (PRISM) as well as the spinal cord injury spasticity evaluation tool (SCI-SET), both established in 2007, are validated and recommended to apply in routine practice. Unfortunately, the SCI-SET is only available in English, Persian and Turkish which hinders the implementation in other language regions.

Therefore the investigators decided to translate and cross-culturally adapt the SCI-SET and create a German version of that questionnaire (SCI-SETde). This finally helps to assess the usefulness of therapeutic interventions and to monitor the course of spasticity in patients. The SCI-SETde will be checked for comprehensibility and tested for cultural aspects in advance to its validation. These are prerequisites that it can later be used in daily routine.

The expected risk and burden for participants is very small because they only have to fill in questionnaires.

The primary objective is to establish the SCI-SETde and to cross-culturally adapt and validate it in a small cohort of patients. The translation and back-translation already happened and the authors of the initial SCI-SET are informed and gave their consent that a German version of this questionnaire may be established.

It is very important that the questionnaire is understandable and well-suited to ask patients about the influence of their spasticity on several areas of daily life. It is necessary to receive feedback on how patients understand each single question and also if any questions are somehow unclear or not enough accurate or specific. To test the validity and reliability of the questionnaire is necessary to evidence its usefulness for assessment.

Test-retest reliability will be assessed by administering the questionnaires two times at the same day and time one week apart. Construct validity will be assessed by comparing the SCI-SETde with scores from additional questionnaires namely, an adapted form of the Penn Spasm Frequency Scale (PSFS) and the self-reported version of the Spinal Cord Independence Measure (SCIM-SR) as well as self-reported impact and severity of spasticity.

There are possible confounders that may interfere with the results. These confounding factors will be assessed on both time points through an additional checklist that asks patients if they suffered from any kind of fracture, decubitus ulcer, any sort of infection, new arisen pain due to any condition as well as any psychogenic trauma.

People within the SCI community of Switzerland will be taken into consideration to participate in this study. The recruitment of the participants will be either a consecutive ongoing recruitment during daily clinical practice or direct contacting of known SCI patients with stated spasticity symptoms. Patients will be informed in detail about the project if they meet all the inclusion criteria and no exclusion criteria is found in routine practice. Participants are not receiving any compensation for their participation in the study. For each patient the project duration is roughly two weeks.

All the data will be stored safely with only authorized people having access to the data corresponding to their duties to manage or analyze the data. The physical data will be entered into the secure databank for final analysis. All data is encoded by giving each participant a unique patient ID that doesn't allow any inference on the identity of the person. The key document with the link between the patient ID and the person behind it will be stored in a secured desk separately from the remaining study documents.

ELIGIBILITY:
Inclusion Criteria:

* SCI for at least six month and presented with spasticity symptoms
* at least 18 years old
* able to understand the instructions as well as the questionnaires
* no expected changes in medical treatment for the duration of the study (~1 month)

Exclusion Criteria:

* inability to provide informed consent
* co-morbidities (e.g. decubitus ulcers, heterotopic ossification, urinary tract infections or other infections) or any psychological state that influences spasticity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Already done in Group description
Sampling Method: Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2021-08-30 (Actual); Primary Completion 2023-01-23 (Actual); Study Completion 2023-01-23 (Actual)

PRIMARY OUTCOMES:
Score of the Spinal Cord Injury - Spasticity Evaluation Tool german version (SCI-SETde) | Two weeks, initial time point and one week later secondary time point
  The score is divided into a negative and a positive subscore as well as a given total overall score resulting from the 35 items which can be rated in the range from (-3) "extremely problematic" to +3 "extremely helpful". So the lowest (negative) achievable score is -105 and indicates a high limitation due to spasticity to execute activities of daily living. The highest achievable score is 105 and indicates a high supporting function of spasticity to execute activities of daily living.
Score from the adapted Penn Spasm Frequency Scale (PSFS) | One day, initial time point
  Frequency score: ranging from 0 "no spasms at all" to 4 "spasms occur more than ten times per hour".
  The score is descriptive indicating the frequency of spasms. The meaning of the score for the outcome remains open because it depends on several factors. If the spasms are beneficiary for example to transfer from wheelchair to car or bed we have to keep in mind that the patient doesn't need to transfer more than ten times per hour. But it might be helpful if the spasms occur several times per hour.
  Intensity score: ranging from 1 "weak" to 3 "strong". The score is descriptive indicating the intensity of spasms. The outcome depends on whether the spasms are limiting or helpful for the patient and depending on whether a strong spasm is more helpful than a moderate spasm. It may be that a strong spasm is limiting whereas a moderate spasm is helpful. So there is no general statement possible and the score can only be interpreted by taking all factors into consideration.
Score from Spinal Cord Independence Measure version 3 self-reported (SCIM III - SR) | One day, initial time point
  The total score of the SCIM III - self reported questionnaire consisting of 19 items.
  Self-care subscale, Items 1-4 (0-20); Respiration and sphincter management subscale, Items 5-8 (0-40); Mobility subscale, Items 9-17 (0-40) Scores are higher in patients that require less assistance or fewer aids to complete basic activities of daily living and life support activities.
Self-evaluation of severity grade of spasticity | One day, initial time point
  The participants are asked to rate the severity grade of their spasticity on a scale ranging from 0 (no spasticity) to 5 (highest imaginable grade of spasticity).
Self-evaluation of limitation in daily life due to spasticity | One day, initial time point
  The participants are asked to rate the extent of limitation in daily life due to their spasticity on a scale ranging from 0 (no limitation) to 5 (highest imaginable limitation).

SECONDARY OUTCOMES:
Asking a question | Two weeks, initial time point and one week later secondary time point
  "Were there any questions that are unclear or undetermined?"
  Response format: Yes/No. "If yes, please indicate which question it concerns and make a suggestion how to write the question."

CONTACTS AND LOCATIONS:
Locations (1):
- Swiss Paraplegic Centre; Centre for pain medicine, Nottwil, Canton of Lucerne, Switzerland

IPD SHARING:
Plan to Share IPD: No